CLINICAL TRIAL: NCT07316283
Title: Effect of Sensorimotor Training Exercises on Shoulder Joint Position Sense Post Mastectomy
Brief Title: Sensorimotor Training Exercises for Shoulder Position Sense
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Huda Tarek Abuassi Mahmoud, Demonstrator at Department of Surgery and Burn - Faculty of Physical Therapy - Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 25698547123654
Record Dates: First submitted 2025-12-17; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Post Mastectomy
Keywords: Sensorimotor training exercises; Shoulder position sense; Post mastectomy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sensorimotor Training Exercises Plus Traditional Physical Therapy Program. (Experimental): Sensorimotor training exercises in addition to the traditional physical therapy program (shoulder ROM exercises, capsular stretching exercises, scapular muscle strengthening exercises, and scapular mobilization) were applied three sessions per week for eight weeks.
  Patients tracked a diagram fixed on the wall using a laser pointer, threw and caught a medicine ball, performed upper-limb weight-bearing exercises on a Swiss ball, and executed wall exercises using a ball. The exercises were performed in three sets of ten repetitions, with one minute of rest between sets, three times per week for eight weeks.
  Traditional physical therapy program included scapular retraction exercises with moderate resistance from standing, shoulder ROM exercises using a shoulder wheel and ladder in flexion and abduction, scapular mobilization from sitting, shoulder Maitland mobilization (inferior, anterior, and posterior glides), and posterior capsule stretching from sitting with two sets of 15 repetitions
  Interventions: Behavioral: Sensorimotor Training Exercises; Behavioral: Traditional Physical Therapy Program
- Traditional Physical Therapy Program (Experimental): Traditional physical therapy program 3 sessions per week for 8 weeks included scapular retraction exercises with moderate resistance from standing, shoulder ROM ex on shoulder wheel and ladder in flexion and abduction, scapular mobilization from sitting, shoulder Mitland mobilization as inferior glide, anterior glide and posterior glide, and posterior capsule stretching from sitting with approximately two sets of 15 repetitions.
  Interventions: Behavioral: Traditional Physical Therapy Program

INTERVENTIONS:
Behavioral: Sensorimotor Training Exercises — Sensorimotor training exercises, in addition to the traditional physical therapy program which included shoulder ROM exercises, capsular stretching exercises, scapular muscle strengthening exercises, and scapular mobilization were applied three sessions per week for eight weeks. Patients tracked a diagram fixed on the wall using a laser pointer, threw and caught a medicine ball, performed upper-limb weight-bearing exercises on a Swiss ball, and executed wall exercises using a ball. Each exercise was performed in three sets of ten repetitions, with one minute of rest between sets. The traditional physical therapy program also included scapular retraction exercises with moderate resistance from standing, shoulder ROM exercises using a shoulder wheel and ladder in flexion and abduction, scapular mobilization from sitting, shoulder Maitland mobilization (inferior, anterior, and posterior glides), and posterior capsule stretching from sitting with two sets of fifteen repetitions.
  Arms: Sensorimotor Training Exercises Plus Traditional Physical Therapy Program.
Behavioral: Traditional Physical Therapy Program — The traditional physical therapy program consisted of scapular retraction exercises with moderate resistance from standing, shoulder range of motion exercises using a shoulder wheel and ladder in flexion and abduction, scapular mobilization from a seated position, shoulder Maitland mobilization including inferior, anterior, and posterior glides, and posterior capsule stretching from a seated position, performed in approximately two sets of fifteen repetitions.

SUMMARY:
Forty-six female patients aged 35-55 years who were suffering from shoulder dysfunction following mastectomy surgeries participated in this study. The participants were recruited from the outpatient clinic of the Faculty of Physical Therapy, Cairo University, and were randomly assigned into two equal groups.

Group A: consisted of 23 patients who received sensorimotor training exercises in addition to a traditional physical therapy program which included shoulder range of motion exercises, capsular stretching exercises, scapular muscle strengthening exercises, shoulder Maitland mobilization, and scapular mobilization.

Group B: consisted of 23 patients who received only the traditional physical therapy program, which included shoulder range of motion exercises, capsular stretching exercises, scapular muscle strengthening exercises, shoulder Maitland mobilization, and scapular mobilization.

Both groups received treatment three sessions per week for a duration of eight weeks.

DETAILED DESCRIPTION:
1. Subjects Forty-six female patients aged 35-55 years who were suffering from shoulder dysfunction following mastectomy surgeries participated in this study. The participants were recruited from the outpatient clinic of the Faculty of Physical Therapy, Cairo University, and were randomly assigned into two equal groups.

   Group A consisted of 23 patients who received sensorimotor training exercises in addition to a traditional physical therapy program, which included shoulder range of motion exercises, capsular stretching exercises, scapular strengthening exercises, scapular mobilization, and shoulder Maitland mobilization. The treatment was administered three sessions per week for eight weeks.

   Group B consisted of 23 patients who received only the traditional physical therapy program, which included shoulder range of motion exercises, capsular stretching exercises, scapular strengthening exercises, scapular mobilization, and shoulder Maitland mobilization. The treatment was administered three sessions per week for eight weeks.
2. Equipment Therapeutic equipment

Sensorimotor training exercises:

Patients performed sensorimotor training exercises that included tracking a diagram fixed on the wall using a laser pointer, throwing and catching a medicine ball, performing upper-limb weight-bearing exercises on a Swiss ball, and executing wall exercises using a ball. The exercises were applied with a dosage of three sets of ten repetitions, with one minute of rest between sets, three times per week for eight weeks.

Traditional physical therapy program:

The traditional physical therapy program was conducted three sessions per week for eight weeks and included scapular retraction exercises with moderate resistance from standing, shoulder range of motion exercises using a shoulder wheel and ladder in flexion and abduction, scapular mobilization from sitting, shoulder Maitland mobilization as inferior, anterior, and posterior glides, and posterior capsule stretching from sitting with approximately two sets of fifteen repetitions.

Measurement equipment

Digital inclinometer:

A digital inclinometer was used as a precise, gravity-based instrument to measure joint angles and range of motion (ROM) with high accuracy. It provided real-time digital readings, making it a reliable and efficient alternative to traditional goniometers. Clinically, it was commonly used to assess joint mobility of the spine, shoulders, hips, and knees, aiding in the evaluation of conditions such as arthritis, ligament injuries, and postoperative stiffness. In addition to ROM assessment, the digital inclinometer was considered a validated tool for evaluating joint position sense (JPS), a key component of proprioception. It was used to measure patients' ability to replicate joint angles, helping to identify neuromuscular control deficits frequently observed in musculoskeletal injuries and post-surgical cases. The objective data obtained supported individualized rehabilitation planning, progress monitoring, and functional recovery. Its portability, ease of use, and high reproducibility made it a valuable instrument in both clinical and research settings.

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* Aged between 35 and 55 years
* Underwent unilateral mastectomy
* Underwent wide local excision
* Underwent axillary dissection
* Presence of shoulder joint dysfunction
* Conscious and able to communicate orally or in writing
* No obvious abnormal spinal morphology or postural abnormalities visible to the naked eye

Exclusion Criteria:

* History of fracture or upper limb surgery within the last 3 months
* History of previous shoulder dislocation or chronic shoulder instability
* Uncontrolled diabetes mellitus
* Inability to communicate effectively or write
* Presence of cognitive, visual, or hearing impairments
* Neurological conditions affecting the upper extremity
* Moderate to severe upper limb lymphedema
* Prior permanent shoulder injury before mastectomy
* Poor physical conditioning or acute pain due to any cause or comorbidity
* Participation in another clinical trial or study that could interfere with the results

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female patients
Enrollment: 46 (Actual)
Dates: Start 2025-09-16 (Actual); Primary Completion 2025-11-16 (Actual); Study Completion 2025-12-16 (Actual)

PRIMARY OUTCOMES:
ShoulderJoint Position Sense | 8 weeks
  A digital inclinometer was used as a validated and reliable tool to assess joint position sense (JPS). It measured the participants' ability to accurately reproduce specific joint angles, providing objective data on proprioceptive accuracy.

CONTACTS AND LOCATIONS:
Overall Officials: Huda Tarek Abuassi, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt